CLINICAL TRIAL: NCT05908097
Title: Enhancing Prospective Thinking in Early Recovery
Brief Title: Enhancing Prospective Thinking in Early Recovery (PARK)
Acronym: PARK
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Brandon G. Oberlin, PhD, Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1805574553; Aims 7-8; PARK (Other: IndianaU); 1R41DA055405-01 (NIH)
Record Dates: First submitted 2023-05-05; First posted 2023-06-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-03

CONDITIONS: Opioid Use; Opioid Use Disorder; Substance Use Disorders
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Two groups: Experimental and Control
Who Masked: Participant
Masking Description: All study participants are randomly assigned to a group prior to study enrollment. Participants will not be made aware of their group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Virtual Reality (Experimental): Participants in this arm will receive the following interventions:
  Virtual Reality Avatar VR plus Treatment As Usual (Intervention)
  Interventions: Device: Virtual Reality Avatar Intervention; Device: Virtual Reality Empty Park
- Sham VR (Control) (Sham Comparator): Participants in this arm will receive the following interventions:
  Sham VR plus Treatment As Usual (Empty Virtual Reality Park)
  Interventions: Device: Virtual Reality Empty Park

INTERVENTIONS:
Device: Virtual Reality Avatar Intervention — In the Virtual Reality Avatar Intervention experience, participants will see an avatar resembling themselves in a park setting.
  Arms: Virtual Reality
Device: Virtual Reality Empty Park — The Virtual Reality Empty Park experience is a habituation experience that does not contain avatars.

SUMMARY:
The goal of this clinical trial is to demonstrate the commercial potential for a novel virtual reality (VR) intervention in preparation for Phase II development. This clinical trial will test the VR intervention for efficacy in reducing opioid use, increasing abstinence, and other self-reported and behavioral focus on future outcomes in individuals in early recovery from opioid use disorder.

* Will the VR group, compared to the control group, have a lower number of opioid use days?
* Will the VR group, compared to the control group, have longer periods of abstinence at the 30-day follow-up?
* Will the VR group, compared to the control group, have significantly increased opioid abstinence rates?
* Will the VR group, compared to baseline and the control group, show increased future self-identification post-VR intervention?
* Will the VR group, compared to baseline and the control group, show increased future orientation post-VR intervention?
* Will the VR group, compared to baseline and the control group, show an increased preference for delayed rewards in a laboratory delay discounting task post-VR intervention?
* Will the VR group, compared to baseline and the control group, exceed in behavioral effects (i.e., future self-identification, future orientation, and increased preference for delayed rewards) at the 30-day follow-up?

Researchers will compare the VR test group and the control group to see if there are differences in the results for the questions outlined above.

ELIGIBILITY:
Inclusion Criteria:

* Abstinence between ≥14 days and ≤ 1 year
* 18-60 years old
* Verbal endorsement of commitment to recovery
* Outpatient
* Psychotropic drugs for SUD-comorbidity
* Mu-Opioid drugs
* Drug/alcohol abstinence ≥ 24 hours at the time of the study day visit
* English comprehension

Exclusion Criteria:

* Unstable medical disorders
* Outside the age range of 18-60
* Habitual drug use
* Smell/taste disorders
* Unstable psychiatric conditions
* Extravagant/elaborate face tattoos

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2025-09-14 (Actual); Study Completion 2025-09-14 (Actual)

PRIMARY OUTCOMES:
Reduced Use of Drug Using Days | Study Day Visit; 30-day Follow-up Visit.
  The VR Avatar experience will change drug using days.
Increased Length of Abstinence | Study Day Visit (Day 1); 30-day Follow-up Visit.
  The VR Avatar experience will change the length of abstinence periods.
Change in Overall Abstinence | Study Day Visit (Day 1); 30-day Follow-up Visit.
  The VR Avatar experience, compared to treatment as usual will change abstinence, measured using a timeline follow-back assessing for substances used from enrollment to study completion.
Future Self-Identification | Study Day Visit (Day 1); 30-day Follow-up Visit
  The VR Avatar Experience will change future self-identification. Future self-identification and change between two time points will also be measured using a proprietary future-self-continuity assessment administered at Study Day Visit (Day 1), and again at the 30-Day Follow-up Visit.
Future Time Orientation | Study Day Visit (Day 1); 30-day Follow-up Visit.
  The Virtual Reality Avatar experience will change orientation toward the future, which will be measured using the Zimbardo Time Perspective Inventory (ZTPI). The ZTPI contains five subscales, and items within each subscale are scored from 1, "very uncharacteristic," to 5, "very characteristic." The subscales are 1) Past-Negative--10 items, higher scores indicative of worse outcomes; 2) Present-Hedonistic--15 items, higher scores indicative of worse outcomes; 3) Future--10 items, higher scores indicative of better outcomes; 4) Past-Positive--9 items, higher scores indicative of better outcomes; and 5) Present-Fatalistic--9 items, higher scores indicative of worse outcomes. Subscales are combined into "future" and "present" categories, then totaled, with higher total scores indicative of worsened outcomes.
Delayed Reward | Study Day Visit (Day 1); 30-day Follow-up Visit.
  The Virtual Reality Avatar experience will change preference for delayed rewards, which will be measured using a behavioral delay discounting task.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon G Oberlin, PhD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - Indiana University School of Medicine - Goodman Hall, Indianapolis, Indiana
  - IUSM - Goodman Hall, Indianapolis, Indiana
  - Serenity Lane Alcohol & Drug Treatment, Coburg, Oregon

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared in accordance with the National Institutes of Health National Data Archive requirements and upon the consent of the study participant.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be shared at the specified submission deadlines assigned by the National Institutes of Health (typically every April or October). Data will be available upon the discretion of the National Institutes of Health.
Access Criteria: No individually identifiable participant data will be submitted to the National Data Archive. All collected participant data is de-identified, and will be made available for other researchers to use upon requests submitted through the National Data Archive portal, and approval from the principal investigator.